CLINICAL TRIAL: NCT02059837
Title: Retrospective Study of Recurrence Patterns Following Conjunctival Autografts for Pterygium Surgery
Brief Title: Clinical Analysis of Recurrence Patterns Following Conjunctival Autografts for Pterygium Surgery
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Hong Kyun Kim, M.D, Kyungpook National University Hospital, Kyungpook National University Hospital
Other Study IDs: KNUH 2014-1
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Recurrent Pterygium
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pterygium,recurrent: Consecutively recorded photographs of recurrent pterygium excision and following grafting were analyzed.
  Interventions: Procedure: recurrent pterygium excision and following grafting

INTERVENTIONS:
Procedure: recurrent pterygium excision and following grafting — The excision of recurrent pterygial tissue and autograft of conjunctiva was done.

SUMMARY:
This study is conducted to evaluate its morphologic reproliferating patterns in patients with pterygium treated with the excision and conjunctival autograft.

DETAILED DESCRIPTION:
The medical records of 116 eyes of 116 patients with pterygium who had pterygium excision and conjunctival autograft between February 2009 and May 2011 were reviewed. Using consecutively recorded photographs, we evaluated preoperative morphologic characteristics and its growth patterns.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent pterygium
* Unilateral or bilateral pterygium
* Both male and female
* Consenting to participate in study

Exclusion Criteria:

* Fibrovascular proliferation secondary to injury
* Severe dry eye syndrome
* Pseudopterygium
* Signs of malignancy on pterygium
* Corneoscleral trauma or corneo-limbal scars

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 116 patients were included. They had pterygium excision and conjunctival autograft surgery and followed by anterior photographs.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Pterygium recurrence pattern | 12 months
  Morphologic recurrence pattern of pterygium using consecutively recorded photographs.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Kyun Kim, M.D., Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Hong Kyun Kim, Daegu, Kyungangpookdo, South Korea

REFERENCES:
- [Derived] Kwon SH, Kim HK. Analysis of recurrence patterns following pterygium surgery with conjunctival autografts. Medicine (Baltimore). 2015 Jan;94(4):e518. doi: 10.1097/MD.0000000000000518. PMID 25634207